CLINICAL TRIAL: NCT01274702
Title: Visual Reconstitution Therapy After Optic Neuritis
Acronym: VISION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Friedemann Paul (Other)
Collaborators: Beuth Hochschule für Technik Berlin (Unknown); NovaVision AG, Zentrum für Sehtherapie (Unknown)
Responsible Party: Sponsor-Investigator, Friedemann Paul, Prof. Dr., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vision Study
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Optic Neuritis; Multiple Sclerosis
Keywords: History of; Patients; acute
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Visual Reconstitution Therapy (Experimental)
  Interventions: Other: Visual Reconstitutions Therapy
- Saccadic Eye Movement Training (Active Comparator)
  Interventions: Other: Saccadic Eye Movement Training

INTERVENTIONS:
Other: Visual Reconstitutions Therapy
  Arms: Visual Reconstitution Therapy
Other: Saccadic Eye Movement Training
  Arms: Saccadic Eye Movement Training

SUMMARY:
Incomplete remission after an optic neuritis attack is not uncommon. Visual reconstitution therapy is a software-based approach that has been shown to substantially improve residual visual field deficits in patients with pre- and postchiasmatic lesions.

The primary hypothesis of this randomized, controlled clinical trial is, that visual reconstitution therapy is superior to active comparator treatment in improving the visual field after optic neuritis.

DETAILED DESCRIPTION:
Patients with an acute optic neuritis (between 60 and 180 days before screening) or with residual visual deficits after a past optic neuritis are randomized in two treatment groups. Group A is instructed to perform software-based visual reconstitution therapy on a home PC daily and regularly for 30 minutes over a period of six month. Group B will perform a similarly, also software-based training program, developed to improve saccadic eye movements rather than visual fields. Patients are blinded to the respective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Definite Optic Neuritis within 60-180 Days or < 12 months before Screening
* Visus > 0.05
* Visus < 0.7 or confirmed visual field deficit
* Ability to give Informed Consent

Exclusion Criteria:

* Systemic Treatment with Glucocorticosteroids within 30 days prior to Screening
* Additional significant ophthalmological disease
* Pregnancy
* History of Epilepsy
* Significant arterial Hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Visual field | 6 months
  visual field perimetry and kampimetry at baseline and after 3 and 6 months

SECONDARY OUTCOMES:
structural retinal changes | 6 months
  Optical coherence Tomography is performe at baselline and after 6 months
Quality of Life | 6 months
  Quality of life is determined by questionaires at baseline and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Paul, MD, Principal Investigator — NeuroCure Clinical Research Center, Charité Universitaetsmedizin Berlin
Locations (1):
- NeuroCure Clinical Reserach Center, Charité Universitaetsmedizin, Berlin, Germany

REFERENCES:
- [Derived] Schinzel J, Schwarzlose L, Dietze H, Bartusch K, Weiss S, Ohlraun S, Paul F, Dorr J. Efficacy of vision restoration therapy after optic neuritis (VISION study): study protocol for a randomized controlled trial. Trials. 2012 Jun 28;13:94. doi: 10.1186/1745-6215-13-94. PMID 22742888
- See also: NeuroCure Clinical Research Center, Charité Berlin, Germany — https://neurocure.de/ncrc/ueber-uns.html